CLINICAL TRIAL: NCT00424333
Title: Efficacy and Safety of Inhaled Compared With Subcutaneous Human Insulin in an Intensive Insulin Regimen for Subjects With Type 1 Diabetes Mellitus: A Six-Month, Outpatient, Parallel Comparative Trial
Brief Title: Six Month Clinical Trial Assessing Efficacy and Safety of Inhaled Insulin in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217-107
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Drug: Inhaled human insulin

SUMMARY:
To determine in subjects with Type 1 Diabetes Mellitus:

1. Whether glycemic control can be achieved at least as effectively with a) an intensive insulin regimen involving pre-meal inhaled insulin plus twice daily subcutaneous NPH insulin as with b) an intensive subcutaneous insulin regimen involving pre-meal regular insulin plus twice daily NPH, given as 4 injections per day. The treatment regimens differ only by the route of delivery of the short acting insulin.
2. The toleration and safety of inhaled insulin therapy and its effects after 6months, if any, on measures of pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes for more than 1 year
* Stable insulin regimen of at least 2 injections per day

Exclusion Criteria:

* Any smoking within the last 6 months. Smoking is not permitted at any time during this study.
* Subjects on insulin pump during 2 months prior to screening.
* Subjects with poorly-controlled asthma, clinically significant chronic obstructive pulmonary disease, or other significant respiratory disease.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320
Dates: Start 1999-05; Study Completion 2000-10

PRIMARY OUTCOMES:
Primary outcome is 24 week change in baseline in HbA1c.

SECONDARY OUTCOMES:
The secondary endpoints include the following efficacy assessments:
Incidence of hypoglycemia
Proportion of subjects with acceptable glycemic control (e.g., HbA1c<8%)
Change from baseline in fasting lipid profile
Change from baseline in fasting plasma glucose level
Change from baseline in meal glucose response (2-hour postprandial increment in plasma glucose)
Dose of insulin (total dose of injected sustained-duration insulin, and total dose of inhaled or injected Regular insulin during the study).
Change from baseline in body weight
Change from baseline in 24-hour home glucose profile (based on the area under the glucose profile curve calculated by the trapezoid rule with special weights assigned to the pre-breakfast and bedtime assessments).
Patient satisfaction and preference.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (30):
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Lutherville, Maryland
  - Pfizer Investigational Site, Waltham, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Charlottsville, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Canada (5):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=107&StudyName=Six+Month+Clinical+Trial+Assessing+Efficacy+and+Safety+of+Inhaled+Insulin+in+Type+1+Diabetes